CLINICAL TRIAL: NCT07270016
Title: Real-Time Engagement for Learning to Effectively Control Type 2 Diabetes: Pilot Study
Brief Title: Pilot-Testing Real-Time Engagement for Learning to Effectively Control Type 2 Diabetes
Acronym: REFLECT2DPilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: San Diego State University (Other); Emory University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Mary Ellen Vajravelu, MD, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY25100193; 1R01DK137803-01A1 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Hyperglycemia; Physical Inactivity; Lifestyle (Sedentary Behavior and Physical Activity); Continuous Glucose Monitoring
Keywords: adolescent; young adult; type 2 diabetes; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm pilot study (Experimental): Participants will engage in pilot-testing a novel smartphone app supporting health behavior change and wear a continuous glucose monitoring device and Fitbit physical activity tracker for 30 days. Questionnaires and interviews will be used to gather participant experiences with the app and device wear.
  Interventions: Other: Healthmine app

INTERVENTIONS:
Other: Healthmine app — Participants will wear study-provided continuous glucose monitoring device and Fitbit physical activity tracker for 30 consecutive days. During the same period, they will use an investigator-developed smartphone app (Healthmine), which is being developed to pair CGM and Fitbit data. Participants will receive up to one message about health behavior change (e.g., physical activity, nutrition) daily and will be able to use Healthmine to log exercise and dietary intake.

SUMMARY:
The goal of this study is to pilot test features of a new smartphone app and to gather feedback related to wearing a continuous glucose monitor (CGM) and a Fitbit device, as well as to obtain input on health behavior-focused messages delivered through the app. The study will enroll English-speaking participants aged 16-24 years who were diagnosed with type 2 diabetes before age 18. Participants will be asked to fill out surveys about diabetes, physical activity, and diet before and after wearing a CGM for 30 days. At the end of wearing the CGM, participants will complete an interview about their experience.

ELIGIBILITY:
Inclusion criteria:

* Ages 16-24 years, any sex or gender
* Diagnosis of type 2 diabetes in childhood (younger than 18 years of age)
* English-speaking (app in English)
* Possession of personal smartphone that is compatible with FreeStyle Libre app

Exclusion Criteria:

• Cognitive impairment or severe psychiatric conditions that could interfere with participation in behavioral intervention for diabetes self-management

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Usability of Healthmine app | 15 days and 30 days after starting study-provided CGM and Healthmine app use
  Assessed via the System Usability Scale (SUS), a 10-item questionnaire measuring perceived usability of a system or technology. Each item is rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"). The total SUS score is calculated by summing the score contributions from each item (for odd-numbered items, subtract 1 from the user response; for even-numbered items, subtract the user response from 5), multiplying the sum by 2.5, resulting in a score ranging from 0 to 100. Higher scores indicate better perceived usability, with scores above 68 considered above average usability.

SECONDARY OUTCOMES:
Days with CGM data | 30-day CGM wear period
  The number of days with continuous glucose monitoring data available will be divided by the total number of requested days of wear (30) to obtain percentage of days with data.
Days with Fitbit data | 30-day Fitbit wear period
  The number of days with Fitbit data available will be divided by the total number of requested days of wear (30) to obtain percentage of days with data.
Mean CGM glucose | 30-day CGM wear period
  Mean glucose obtained from study-provided CGM
Step count | 30-day Fitbit wear period
  Step count data will be obtained via study-provided Fitbit.
Diabetes Self-Management | Baseline and 30 days (change from baseline to 30 days)
  Assessed via the Diabetes Self-Management Questionnaire (DSMQ), a 16-item self-report questionnaire measuring diabetes self-care activities associated with glycemic control. Each item is rated on a 4-point Likert scale (0 = "does not apply to me" to 3 = "applies to me very much"). Items are summed (after reverse-coding negatively worded items) and transformed to a 0-10 scale, where higher scores indicate better self-management.
Treatment Self-Regulation | Baseline and 30 days (change from baseline to 30 days)
  Assessed via the Treatment Self-Regulation Questionnaire (TSRQ), a questionnaire measuring the degree to which a person's motivation for health behaviors is relatively autonomous (self-determined) versus controlled (motivated by external factors). Items are rated on a 7-point Likert scale (1 = "not at all true" to 7 = "very true"). The TSRQ yields subscale scores for autonomous regulation, controlled regulation, and amotivation, with higher scores on each subscale indicating greater levels of that type of motivation.
Self-Reported Physical Activity | Baseline and 30 days (change from baseline to 30 days)
  Assessed via the PACE+ Physical Activity Measure, a brief self-report questionnaire measuring physical activity levels. Participants report the number of days per week they engage in moderate or vigorous physical activity for at least 30 minutes (or 60 minutes for adolescents). The measure yields separate scores for moderate and vigorous activity (each ranging from 0-7 days per week), with higher scores indicating greater physical activity frequency.
Diet Quality | Baseline and 30 days (change from baseline to 30 days)
  Assessed via the Prime Diet Quality Score (PDQS), a food-based dietary assessment tool that evaluates diet quality across 15 food group components. The PDQS includes 10 adequacy components (dark green leafy vegetables, cruciferous vegetables, carrots, other vegetables, citrus fruits, other fruits, fish/seafood, eggs, whole grains, and low-fat dairy) and 5 moderation components (red meat as main dish, processed meat, refined grains and baked goods, sugar-sweetened beverages, and fried foods). Each component is scored based on consumption frequency, with higher scores indicating greater intake of health-promoting foods and lower intake of foods that should be consumed in moderation. The total PDQS ranges from 0-30, with higher scores indicating better overall diet quality.
Glucose monitoring satisfaction | 30 days (following CGM wear period)
  Assessed via the Glucose Monitoring Satisfaction Survey (GMSS) for Type 2 Diabetes, a 15-item questionnaire measuring patient satisfaction with their glucose monitoring device. Items are rated on a 5-point Likert scale (1 = "strongly disagree" to 5 = "strongly agree"). The GMSS yields four subscale scores: Openness (items 1, 8, 10, 14), Emotional Burden (items 2, 5, 9, 13), Behavioral Burden (items 3, 6, 11, 15), and Worthwhileness (items 4, 7 [reverse coded], 12). Subscale scores are calculated as the mean of item responses, with higher scores indicating greater openness, greater burden (for burden subscales), and greater worthwhileness, respectively. A total satisfaction score is calculated as the mean of all items after reverse-coding items 2, 3, 5, 6, 7, 9, 11, 13, and 15, with higher total scores indicating greater overall satisfaction with glucose monitoring.
Glucose coefficient of variation | 30-day CGM wear period
  Based on CGM glucoses, coefficient of variation will be calculated by dividing the standard deviation of glucose readings by the mean glucose level, then multiplying by 100 to get a percentage.
Glucose time below range | 30-day CGM wear period
  Percent of time with CGM glucose less than 70 mg/dL
Glucose time in range | 30-day CGM wear period
  Percent of time with CGM glucose 70-180 mg/dL
Glucose time above range | 30-day CGM wear period
  Percent of time with CGM glucose above 180 mg/dL
Mean amplitude of glycemic excursions | 30-day CGM wear period
  A measure of glucose variability calculated from CGM data, calculated by dividing the standard deviation of glucose readings by the mean glucose level, then multiplying by 100 to get a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Vajravelu, MD, MSHP, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No